CLINICAL TRIAL: NCT03869645
Title: CAPERE Thrombectomy System Post-Market Clinical Follow Up Study
Status: Terminated | Type: Observational
Why Stopped: Change in Sponsor
Sponsor: Medtronic Endovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: TP18-0009
Record Dates: First submitted 2019-03-07; First posted 2019-03-11 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Observational Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: CAPERE Thrombectomy System — Mechanical thrombectomy of acute thrombus in peripheral vasculature with the CAPERE Thrombectomy System

SUMMARY:
A prospective, single-arm, non-blinded study, intending to collect and evaluate data in up to forty (40) human subjects with acute thrombosis, treated with the CAPERE™ Thrombectomy System.

DETAILED DESCRIPTION:
A prospective, single-arm, non-blinded study, intending to collect and evaluate data in up to forty (40) human subjects with acute thrombosis, treated with the CAPERE™ Thrombectomy System.

Subjects will be evaluated based on VEINES QoL survey pre- and post-treatment (30-days).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are greater than or equal to 18 years of age
* Patients with clinical signs, symptoms and presentation consistent with acute thrombosis; onset of symptoms < 14 days
* Patients cleared medically for invasive endovenous procedures

Exclusion Criteria:

* Patients with IVC filter in area to be treated
* Patients who are < 18 years of age.
* Known anaphylactic reaction of radiographic contrast agents that cannot be pre- treated
* Imaging evidence or other evidence that suggests the participant is not appropriate for mechanical thrombectomy intervention
* Female who is pregnant or nursing
* Concurrent participation in another investigational drug or device treatment study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with clinical symptoms of extremity swelling with ultrasound evidence of acute thrombosis in the peripheral vasculature.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
Restoration of blood flow | Day 0 - Intervention
  Clearance of clot and restoration of venous flow of the affected vessel as confirmed using venogram immediately post-procedure

SECONDARY OUTCOMES:
Device Success | Day 0
  Successful withdrawal of device along with clots without clinically significant emboli, permanent vessel trauma, entry site aneurysm, major bleeding complications
Technical Success Rate | Day 0
  Ratio of successful thrombus removals and total number of participants
Thrombus removal rate | Day 0
  percent of thrombus removal comparing pre-treatment to post-treatment venography
VEINES Survey | </= Day 0 and Day 30
  Evaluation of quality of life (QoL) before and after treatment based on VEINES survey responses. Eight (8) QoL questions related to the patient's leg problems are evaluated and their scores aggregated into a single QoL score. The resultant aggregated QoL range is from 26 - 108 where the higher the number the higher the quality of life.
Safety Endpoint | 30 days
  Evaluation of the incidence of unanticipated adverse device events: estimated to be less than or equal to 5%

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Wu, MD, Principal Investigator — Unity Health Toronto
Locations (3):
- United States (3):
  - Memorial Health Services, Fountain Valley, California
  - St. Joseph Hospital, Orange, California
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No